CLINICAL TRIAL: NCT02174679
Title: 68Ga-DOTATATE Imaging in Neuroendocrine Tumors
Brief Title: 68Ga DOTATATE PET/CT in Neuroendocrine Tumors (Expanded Access)
Status: No longer available | Type: Expanded Access
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: DOTATATE12-001920EA; NCI-2016-01796 (Other: CTRP); JCCCID324 (Other: Jonsson Comprehensive Cancer Center)
Record Dates: First submitted 2014-06-20; First posted 2014-06-25 (Estimated); Last update posted 2020-07-27 (Actual); Status verified 2019-05

CONDITIONS: Carcinoid Cancer; Neuroendocrine Tumors; Medullary Thyroid Cancer; Cancers Expressing Somatostatin Receptors
MeSH Terms: conditions — Neuroendocrine Tumors; Carcinoma, Medullary | interventions — Ga(III)-DOTATOC

INTERVENTIONS:
Drug: 68Ga DOTATATE — Patients with somatostatin receptor positive tumors will be evaluated with 68Ga-DOTATATE PET/CT.
  Other Names: 68Ga DOTATATE PET/CT Scan

SUMMARY:
To evaluate 68Ga-DOTATATE PET/CT for staging of patients with carcinoid, neuroendocrine tumors, medullary thyroid cancer and other cancers expressing somatostatin receptors.

DETAILED DESCRIPTION:
This is an expanded access study with a total of 300 participants with NET and suspected SSTR positive tumors. Eligible participants will undergo baseline assessments at enrollment. Study participants will receive 68Ga-DOTATATE and will undergo a PET/CT imaging study. All patients referred by Oncologists will be screened by a UCLA Nuclear Medicine physician and then accepted for scanning if clinically appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years the time of radiotracer administration
* Provides written informed consent
* Known diagnosis of NET or suspected SSTR positive tumors Women of childbearing age must have a negative pregnancy test at screening/baseline
* Able to remain still for duration of each imaging procedure (about 30 minutes)

Exclusion Criteria:

* Less than 18 years-old at the time of radiotracer administration
* Pregnant or nursing
* Inability to complete the needed investigational and standard-of-care imaging examinations due to other reasons (severe claustrophobia, radiation phobia, etc.)
* Any additional medical condition, serious concurrent illness, or other extenuating circumstance that, in the opinion of the Investigator, may significantly interfere with study compliance.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Czernin, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Hospital, Los Angeles, California, United States

REFERENCES:
- [Background] Modlin IM, Kidd M, Hinoue T, Lye KD, Murren J, Argiris A. Molecular strategies and 111in-labelled somatostatin analogues in defining the management of neuroendocrine tumour disease: a new paradigm for surgical management. Surgeon. 2003 Jun;1(3):137-43. doi: 10.1016/s1479-666x(03)80092-6. PMID 15570748
- [Background] Modlin IM, Latich I, Zikusoka M, Kidd M, Eick G, Chan AK. Gastrointestinal carcinoids: the evolution of diagnostic strategies. J Clin Gastroenterol. 2006 Aug;40(7):572-82. doi: 10.1097/00004836-200608000-00003. PMID 16917396
- [Background] Graham MM, Menda Y. Radiopeptide imaging and therapy in the United States. J Nucl Med. 2011 Dec;52 Suppl 2:56S-63S. doi: 10.2967/jnumed.110.085746. PMID 22144556
- [Background] Virgolini I, Ambrosini V, Bomanji JB, Baum RP, Fanti S, Gabriel M, Papathanasiou ND, Pepe G, Oyen W, De Cristoforo C, Chiti A. Procedure guidelines for PET/CT tumour imaging with 68Ga-DOTA-conjugated peptides: 68Ga-DOTA-TOC, 68Ga-DOTA-NOC, 68Ga-DOTA-TATE. Eur J Nucl Med Mol Imaging. 2010 Oct;37(10):2004-10. doi: 10.1007/s00259-010-1512-3. PMID 20596866
- [Background] Buchmann I, Henze M, Engelbrecht S, Eisenhut M, Runz A, Schafer M, Schilling T, Haufe S, Herrmann T, Haberkorn U. Comparison of 68Ga-DOTATOC PET and 111In-DTPAOC (Octreoscan) SPECT in patients with neuroendocrine tumours. Eur J Nucl Med Mol Imaging. 2007 Oct;34(10):1617-26. doi: 10.1007/s00259-007-0450-1. Epub 2007 May 23. PMID 17520251
- [Derived] Calais J, Czernin J, Eiber M, Fendler WP, Gartmann J, Heaney AP, Hendifar AE, Pisegna JR, Hecht JR, Wolin EM, Slavik R, Gupta P, Quon A, Schiepers C, Allen-Auerbach MS, Herrmann K. Most of the Intended Management Changes After 68Ga-DOTATATE PET/CT Are Implemented. J Nucl Med. 2017 Nov;58(11):1793-1796. doi: 10.2967/jnumed.117.192450. Epub 2017 May 4. PMID 28473600
- See also: UCLA Ahmanson Translational Imaging Division — http://pet.ucla.edu